CLINICAL TRIAL: NCT04600414
Title: Collaborating to Heal Addiction and Mental Health in Primary Care
Acronym: CHAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Arkansas (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, John Cooper Fortney, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SITE00000376; UF1MH121942 (NIH)
Record Dates: First submitted 2020-10-09; First posted 2020-10-23 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Opioid-use Disorder; Mental Health Disorder
Keywords: Primary Care; Collaborative Care
MeSH Terms: conditions — Opioid-Related Disorders; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial. Clinics within healthcare systems are paired and randomized to intervention or control.
Who Masked: Outcomes Assessor
Masking Description: Outcomes are assessed by patient survey, and survey administrators will be masked to randomizations status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care for Mental Health Symptoms (Active Comparator): Collaborative Care Management is an integrated care model that operationalizes the principles of the chronic care model to improve access to evidence-based treatments for mental health disorders.
  Interventions: Other: Collaborative Care for Mental Health Symptoms
- Collaborative Care for Opioid Use Disorder and Mental Health Symptoms (Experimental): Collaborative Care Management is an integrated care model that operationalizes the principles of the chronic care model to improve access to evidence-based treatments for opioid use disorder.
  Interventions: Other: Collaborative Care for Mental Health Symptoms; Other: Collaborative Care for Opioid Use Disorder and Mental Health Symptoms

INTERVENTIONS:
Other: Collaborative Care for Mental Health Symptoms — CoCM is based on six key principles: 1) evidence-based, 2) measurement-based, 3) team-based, 4) population-based, 5) patient-centered, and 6) accountable. CoCM supports the delivery of evidence-based pharmacological and psychosocial treatments. CoCM is measurement-based with screening and monitoring of patient-reported outcomes over time to assess treatment response and facilitate treatment adjustments. CoCM is team-based led by a primary care provider with support from a care manager in consultation with a psychiatrist who provides treatment recommendations for patients who are not responding. CoCM is population-based whereby a registry is used to monitor treatment engagement and facilitate the identification of patients falling through the cracks. CoCM is patient-centered with proactive outreach to engage and activate patients. Collaborative care is accountable with continuous quality improvement to meet clinic performance benchmarks.
Other: Collaborative Care for Opioid Use Disorder and Mental Health Symptoms — Pharmacologic treatment of OUD will rely mainly on transmucosal buprenorphine/naloxone prescribed by primary care providers with DATA 2000 waivers. Measurement-based care and "treat to target" are fundamental principles of CoCM and will be incorporated into the intervention. Care managers will ask four yes/no questions about: 1) opioid withdrawal symptoms, 2) illicit opioid craving, 3) illicit opioid use, 4) medication side effects. If necessary, consulting psychiatrists will then recommend a change to the treatment plan to the primary care provider. In the case of buprenorphine/naloxone, options for changing the treatment plan include: 1) increasing the dosage (max dose 32mg), 2) augmenting with clonidine, 3) switching to injectable buprenorphine, and/or 4) intensifying psychosocial interventions. If the patient is experiencing medication side effects, but not opioid withdrawal symptoms or illicit opioid craving, consideration will be given to lowering the medication dosage.
  Arms: Collaborative Care for Opioid Use Disorder and Mental Health Symptoms

SUMMARY:
The gold-standard intervention for Opioid Use Disorder (OUD) is Medication for Opioid Use Disorder (MOUD). Because more patients with OUD need access to MOUD in primary care, the investigators are testing whether the Collaborative Care model (CoCM) is effective at treating both mental health disorders (MHD) and OUD concurrently in primary care settings. The intervention is CoCM for MHD and OUD. The active control is CoCM for MHD, but not treating OUD. The primary objective is to compare patient-reported outcomes in the intervention and control groups, and will be tested with in an Effectiveness trial. The secondary objective is to compare the detection of OUD pre- versus post-OUD screening implementation, and will be tested using a Pre-Post trial design. The exploratory objective is to compare intervention clinics randomized to a low-intensity sustainability implementation strategy or a high-intensity sustainability strategy, and will be tested in an Implementation trial.

DETAILED DESCRIPTION:
This multi-site study involves a sequence of trials (Pre-Post -> Effectiveness -> Implementation 3) to examine our primary, secondary and exploratory objectives.

1. Pre-Post trial (secondary objective) - Screening for Opioid User Disorder (OUD) will be integrated into Mental Health Disorder (MHD) screening and electronic health record (EHR) data will be used to determine if screening improves the detection of new cases of OUD during the first six months of the trial compared to the six months prior.
2. Cluster randomized Effectiveness trial (primary objective) - The primary objective of the trial is to test the effectiveness of delivering (Medication for OUD) MOUD in the context of Collaborative Care Management (CoCM) for MHD, hereafter termed the "intervention" compared to CoCM for MHD only hereafter termed the "control". All 24 sites have previously partnered with the AIMS Center to implement CoCM for MHD. After monitoring CoCM for MHD fidelity during a three month "run in" phase, the investigators will categorize clinics into one of two cohorts and then randomize them.

   * Cohort 1 (n=600) - Randomize clinics with high CoCM for MHD fidelity to sequentially adding MOUD for OUD (intervention group) or maintenance CoCM for MHD only (control group).
   * Cohort 2 (n=600) - Randomize clinics with low CoCM for MHD fidelity to simultaneous implementation of CoCM for MHD and OUD (intervention group ) or CoCM for MHD only (control group).
3. Cluster randomized Implementation trial (exploratory objective) - At the end of the Effectiveness trial, the intervention clinics will be randomized to receive a low-intensity or high-intensity implementation strategy to promote sustainability

ELIGIBILITY:
Inclusion Criteria:

1. Screen positive on the NIDA-ASSIST OUD items or referred to the trial by one of the clinic's providers AND
2. Meet clinical criteria for ≥2 symptoms of OUD on the DSM-5 checklist (administered by a clinician) AND
3. Screen positive for depression on the PHQ-9 (≥ 5) OR generalized anxiety on the GAD-7 (≥ 5) OR PTSD on the PC-PTSD-5 (≥ 1) within past 6 months.

Exclusion Criteria:

1. Patient is being prescribed psychotropic medication (including MOUD) by a Mental Health Care Specialist (typically practicing in a specialty addiction treatment setting).
2. Patient is receiving or prefers to seek OUD treatment in specialty care setting including opioid treatment programs
3. Patient does not speak English or Spanish
4. Patient is younger than 18 years of age
5. Patient has a diagnosis of dementia
6. Patient lacks the capacity to provide informed consent
7. Patient doesn't plan on getting care at the clinic for the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fortney, PhD, Principal Investigator — University of Washington
Locations (33):
- United States (33):
  - Unity Health Care Minnesota Avenue Health Center, Washington D.C., District of Columbia
  - Unity Health Care Anacostia Health Center, Washington D.C., District of Columbia
  - Emory University Hospital Midtown-Radiology, Atlanta, Georgia
  - Emory Clinic at Saint Joseph's - Primary Care, Atlanta, Georgia
  - Emory at Dunwoody - Family Medicine, Dunwoody, Georgia
  - Emory at Rockbridge - Primary Care & Nephrology, Stone Mountain, Georgia
  - Kootenai Clinic Family Medicine Ironwood, Coeur d'Alene, Idaho
  - Kootenai Clinic Family Medicine Residency, Coeur d'Alene, Idaho
  - Kootenai Clinic Internal Medicine Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Family Medicine Post Falls, Post Falls, Idaho
  - Minooka Healthcare Center - Ridge Road Campus, Channahon, Illinois
  - Oak Street Health Madison St., Chicago, Illinois
  - Oak Street Health Hermosa, Chicago, Illinois
  - Gardner Healthcare Center of Morris Hospital, Gardner, Illinois
  - Minooka Healthcare Center of Morris Hospital - Mondamin St., Minooka, Illinois
  - Morris Healthcare Center of Morris Hospital - Dresden Drive, Morris, Illinois
  - Oak Street Health Chicago Ave Primary Care Clinic, Oak Park, Illinois
  - Oak Street Health Gary Primary Care Clinic, Gary, Indiana
  - Beth Israel Lahey Health Primary Care & Specialty Care, Beverly Medical Associates, Beverly, Massachusetts
  - Beth Israel Deaconess HealthCare-Chelsea, Chelsea, Massachusetts
  - Berkshire Hillcrest Family Health Center, Pittsfield, Massachusetts
  - Berkshire Williamstown Medical, Williamstown, Massachusetts
  - OneWorld Community Health Centers Livestock Exchange, Omaha, Nebraska
  - OneWorld Community Health Centers Northwest, Omaha, Nebraska
  - Oak Street Health Pleasant Grove Primary Care Clinic, Dallas, Texas
  - Oak Street Health Meadowbrook Primary Care Clinic, Fort Worth, Texas
  - Oak Street Health North Side Primary Care, Fort Worth, Texas
  - Northshore Medical Group Stevenson, Stevenson, Washington
  - PeaceHealth Family Medicine of Southwest Washington, Vancouver, Washington
  - Peace Health Fisher's Landing, Vancouver, Washington
  - Northshore Medical Group White Salmon, White Salmon, Washington
  - UW Health Yahara Clinic, Monona, Wisconsin
  - UW Health Deforest-Windsor Clinic, Windsor, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The PIs will follow the NIH Healthcare Systems Research Collaboratory recommendations for data sharing. Data from this project will be made as widely and freely available as possible while safeguarding the privacy of participants, and protecting confidential and proprietary data. Data will be shared via the National Database for Clinical Trials (NDCT) related to Mental Illness. Investigators will certify the quality of all data generated by grants funded under this FOA prior to submission to NDCT and review their data for accuracy after submission. Precautions will be made regarding patient confidentiality, including HIPAA-compliant patient de-identification for all patients. Public-use datasets will not include patient identifiers, or health system identifiers, characteristics or prescribing/referral practices of individual providers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available in May of 2024.

REFERENCES:
- [Derived] Fortney JC, Ratzliff AD, Blanchard BE, Ferro L, Chase E, Rouvere J, Duncan MH, Merrill JO, Simpson T, Williams EC, Austin EJ, Curran GM, Schoenbaum M, Heagerty PJ, Saxon AJ. Collaborative Care for Opioid Use Disorder in Primary Care: A Hybrid Type 2 Cluster Randomized Clinical Trial. JAMA Psychiatry. 2025 Oct 1;82(10):956-966. doi: 10.1001/jamapsychiatry.2025.2126. PMID 40833733

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinics
Groups:
- Control - Collaborative Care for Mental Health Symptoms: Collaborative Care Management is an integrated care model that operationalizes the principles of the chronic care model to improve access to evidence-based treatments for mental health conditions.
  Collaborative Care (CoCM) is based on six key principles: 1) evidence-based, 2) measurement-based, 3) team-based, 4) population-based, 5) patient-centered, and 6) accountable. CoCM supports the delivery of evidence-based pharmacological and psychosocial treatments. CoCM is measurement-based with screening and monitoring of patient-reported outcomes over time to assess treatment response and facilitate treatment adjustments. CoCM is team-based led by a primary care provider with support from a care manager in consultation with a psychiatrist who provides treatment recommendations for patients who are not responding. CoCM is population-based whereby a registry is used to monitor treatment engagement and facilitate the identification of patients falling through the cracks. CoCM is patient-centered with proactive outreach to engage and activate patients. Collaborative care is accountable with continuous quality improvement to meet clinic performance benchmarks.
- Intervention - Collaborative Care for Opioid Use Disorder and Mental Health Symptoms: Collaborative Care Management is an integrated care model that operationalizes the principles of the chronic care model to improve access to evidence-based treatments for mental health conditions and opioid use disorder.
  Collaborative Care for Opioid Use Disorder: Pharmacologic treatment of OUD will rely mainly on transmucosal buprenorphine/naloxone prescribed by primary care providers with DATA 2000 waivers. Measurement-based care and "treat to target" are fundamental principles of CoCM and will be incorporated into the intervention. Care managers will ask four yes/no questions about: 1) opioid withdrawal symptoms, 2) illicit opioid craving, 3) illicit opioid use, 4) medication side effects. If necessary, consulting psychiatrists will then recommend a change to the treatment plan to the primary care provider. In the case of buprenorphine/naloxone, options for changing the treatment plan include: 1) increasing the dosage (max dose 32mg), 2) augmenting with clonidine, 3) switching to injectable buprenorphine, and/or 4) intensifying psychosocial interventions. If the patient is experiencing medication side effects, but not opioid withdrawal symptoms or illicit opioid craving, consideration will be given to lowering the medication dosage.
Period: Overall Study
Arm/Group | Control - Collaborative Care for Mental Health Symptoms | Intervention - Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Started | 144; 17 Clinics | 110; 17 Clinics
Completed | 115; 16 Clinics | 84; 16 Clinics
Not Completed | 29; 1 Clinics | 26; 1 Clinics

BASELINE CHARACTERISTICS:
Population: Not all enrolled patients completed the baseline survey.
Groups:
- Collaborative Care for Mental Health Symptoms: Collaborative Care Management is an integrated care model that operationalizes the principles of the chronic care model to improve access to evidence-based treatments for mental health conditions.
  Collaborative Care (CoCM) is based on six key principles: 1) evidence-based, 2) measurement-based, 3) team-based, 4) population-based, 5) patient-centered, and 6) accountable. CoCM supports the delivery of evidence-based pharmacological and psychosocial treatments. CoCM is measurement-based with screening and monitoring of patient-reported outcomes over time to assess treatment response and facilitate treatment adjustments. CoCM is team-based led by a primary care provider with support from a care manager in consultation with a psychiatrist who provides treatment recommendations for patients who are not responding. CoCM is population-based whereby a registry is used to monitor treatment engagement and facilitate the identification of patients falling through the cracks. CoCM is patient-centered with proactive outreach to engage and activate patients. Collaborative care is accountable with continuous quality improvement to meet clinic performance benchmarks.
- Collaborative Care for Opioid Use Disorder and Mental Health Symptoms: Collaborative Care Management is an integrated care model that operationalizes the principles of the chronic care model to improve access to evidence-based treatments for mental health conditions and opioid use disorder.
  Collaborative Care for Opioid Use Disorder: Pharmacologic treatment of OUD will rely mainly on transmucosal buprenorphine/naloxone prescribed by primary care providers with DATA 2000 waivers. Measurement-based care and "treat to target" are fundamental principles of CoCM and will be incorporated into the intervention. Care managers will ask four yes/no questions about: 1) opioid withdrawal symptoms, 2) illicit opioid craving, 3) illicit opioid use, 4) medication side effects. If necessary, consulting psychiatrists will then recommend a change to the treatment plan to the primary care provider. In the case of buprenorphine/naloxone, options for changing the treatment plan include: 1) increasing the dosage (max dose 32mg), 2) augmenting with clonidine, 3) switching to injectable buprenorphine, and/or 4) intensifying psychosocial interventions. If the patient is experiencing medication side effects, but not opioid withdrawal symptoms or illicit opioid craving, consideration will be given to lowering the medication dosage.
- Total: Total of all reporting groups
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms | Total
Number analyzed (Participants) | 132 | 100 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.3) | 39.1 (12.3) | 40.9 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 57 | 35 | 92
  Woman | 74 | 65 | 139
  Non-binary or gender fluid | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 122 | 89 | 211
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 5 | 15
  White | 112 | 81 | 193
  More than one race | 7 | 7 | 14
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 132 | 100 | 232
Opioid Use Other Than As Prescribed [Mean (Standard Deviation); unit: Days] | 5.73 (10.79) | 3.66 (8.27) | 4.84 (9.70)
Mental Health Functioning [Mean (Standard Deviation); unit: units on a scale] | 34.18 (13.48) | 34.81 (12.77) | 34.45 (13.17)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use Other Than As Prescribed
Description: Illicit opioid use will be measured from self-report using Opioid use will be measured using item 7E from the Brief Addiction Monitor (BAM) with the following preamble: "The next question asks about your use of street opioids and use of prescription opioids that were not prescribed to you by a healthcare provider. In the past 30 days, how many days did you use opiates such as Heroin, Morphine, Dilaudid, Demerol, Oxycontin, oxy, codeine (e.g., Tylenol 2,3,4), Percocet, Vicodin, Fentanyl, etc.? Do not count times you used buprenorphine, suboxone, or methadone as directed by a healthcare provider."
Time Frame: 6 months
Population: Participants completing the 6-month follow-up survey.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Number analyzed (Participants) | 118 | 85
Days | 3.92 (8.86) | 0.72 (3.61)
Statistical Analysis 1: Comparison: Collaborative Care for Mental Health Symptoms vs Collaborative Care for Opioid Use Disorder and Mental Health Symptoms; Test type: Superiority; p < 0.001, Multi-level model to account for cluster; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0.03 to 0.38]

2. Primary Outcome: Mental Health Functioning
Description: Mental health functioning will be measured from self-report using the Mental Health Component Summary Score from the SF12V (range 0-100, higher scores are better)
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Number analyzed (Participants) | 118 | 85
units on a scale | 38.90 (13.20) | 39.09 (14.03)
Statistical Analysis 1: Comparison: Collaborative Care for Mental Health Symptoms vs Collaborative Care for Opioid Use Disorder and Mental Health Symptoms; Test type: Superiority; p = 0.532, Multi-level model to account for cluster; Mean Difference (Final Values) = -1.20, 95% CI 2-sided [-4.97 to 2.57]

3. Secondary Outcome: Depression Symptoms
Description: Depression symptoms will be measured from self report using the SCL-20 (range 0-4, higher scores are worse)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Number analyzed (Participants) | 118 | 85
units on a scale | 1.30 (0.82) | 1.24 (0.83)

4. Secondary Outcome: Anxiety Symptoms
Description: Anxiety symptoms will be measured from self report using the PROMIS Measure - Emotional Distress, Anxiety, Short Form 7a (range 0-100, higher scores are worse)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Number analyzed (Participants) | 118 | 85
units on a scale | 55.61 (7.85) | 55.82 (7.72)

5. Secondary Outcome: PTSD Symptoms
Description: PTSD symptoms will be measured from self-report using the PCL-5 (range 0-80, higher scores are worse)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Number analyzed (Participants) | 118 | 85
units on a scale | 28.29 (19.01) | 27.32 (18.21)

6. Secondary Outcome: Medications for Opioid Use Disorder (MOUD) Persistence
Description: MOUD persistence will be measured from self report and specified as the proportion of days the study participant reported taking the MOUD medication during the 90 prior to the 6-month follow-up.
Time Frame: 90 days prior to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: proportion
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Number analyzed (Participants) | 115 | 84
proportion | 0.74 (0.42) | 0.90 (0.29)

7. Other Pre Specified Outcome: Perceived Access to Addiction Care for Opioid Use Disorder
Description: Perceived access to care will be measured from self report using the Assessment of Perceived Access to Care (APAC) instrument (range 1-5, higher scores are better)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Number analyzed (Participants) | 118 | 85
units on a scale | 3.82 (0.86) | 4.00 (0.74)

8. Other Pre Specified Outcome: Risk Factors for Premature Mortality
Description: Risk factors will include self-reported intent on self-harm, self-reported overdose, self-reported discontinuation of medications for opioid use disorder and the following adverse events reports: overdose, suicide attempt, hospitalization and ER admission.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Count of risk factors for mortality
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
Number analyzed (Participants) | 118 | 85
Count of risk factors for mortality | 0.51 (0.50) | 0.34 (0.47)

ADVERSE EVENTS:
Time Frame: Baseline - 6 month follow-up
Arm/Group | Collaborative Care for Mental Health Symptoms | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms
All-Cause Mortality (participants affected / at risk) | 1/132 | 0/100
Serious Adverse Events (participants affected / at risk) | 16/132 | 14/100
Other Adverse Events (participants affected / at risk) | 1/132 | 3/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collaborative Care for Mental Health Symptoms (N=132) | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms (N=100)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Non-lethal overdose (that resulted in hospitalization or ED visit) (Psychiatric disorders) | 5 (6) | 2 (3)
Hospitalization (not related to suicide or NSSI - not including non-lethal overdose) (General disorders) | 4 (4) | 1 (6)
Hospitalization (related to suicide or NSSI - not including non-lethal overdose) (Psychiatric disorders) | 1 (1) | 1 (1)
ED visit (not due to suicide attempt or NSSI- not including non-lethal overdose) (General disorders) | 9 (22) | 12 (24)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collaborative Care for Mental Health Symptoms (N=132) | Collaborative Care for Opioid Use Disorder and Mental Health Symptoms (N=100)
Various ailments or injuries not resulting in hospitalization or ED visit (General disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT04600414/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT04600414/SAP_001.pdf